CLINICAL TRIAL: NCT01921556
Title: The Improving Care in Chronic Obstructive Lung Disease Study: CAROL Improving Processes of Care and Quality of Life of COPD Patients in Primary Care: A Cluster Randomized Trial
Brief Title: The Improving Care in Chronic Obstructive Lung Disease Study A Cluster Randomized Trial
Acronym: CAROL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CAROL
Record Dates: First submitted 2013-07-30; First posted 2013-08-13 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- QualiCCare education (Active Comparator): "QualiCCare"education is a training workshop designed to educate professionals on the guidelines but also and particularly governing professional behavior by feedback, reminders and pathways that help to change their attitudes and care behavior. Based on behavioral and learning theory, QualiCCare intervention not only tries to increase knowledge but also internal motivation and decision making by stimuli and resources and by written instruments that guide evidence based decision support.
  Interventions: Behavioral: active comparator, QualiCCare education
- usual care (No Intervention): The practices randomized to the control group apply care as usual

INTERVENTIONS:
Behavioral: active comparator, QualiCCare education — Physicians randomized into the intervention group get a "QualiCCare" training workshop designed to educate professionals on the guidelines but also and particularly governing professional behavior by feedback, reminders and pathways that help to change their attitudes and care behavior. Based on behavioral and learning theory, QualiCCare intervention not only tries to increase knowledge but also internal motivation and decision making by stimuli and resources and by written instruments that guide evidence based decision support.
  Arms: QualiCCare education

SUMMARY:
Background The Swiss health ministry launched a national quality program "QualiCCare" in 2011 to improve healthcare for patients with COPD.

The aim of this study is to determine whether participation in the COPD quality initiative ("QualiCCare") improves adherence to recommended clinical processes and shows impact on patients COPD care and on quality of life in patients with COPD.

DETAILED DESCRIPTION:
The care in obstructive lung disease study (CAROL) is a cluster-randomized controlled trial with randomization on the practice level. Thirty practices will be randomly assigned to equally sized intervention group or control group.

Each General Practioner (GP) of a practice will approach consecutively and regardless the reason for the current encounter, COPD patients diagnosed by spirometric evaluation (FEV1/ FVC < 0.70), aged 45 years older, with a smoking history of = 10 pack-years (PY). GPs in the intervention group will receive "QualiCCare" education, which addresses knowledge, decision-making and behavioural aspects as well as delivery of care according to COPD quality indicators and evidence based key elements. In the control group no educational intervention will be applied and COPD patients will be treated as usual. The study period is one year.

The primary outcome measure is an aggregated score of relevant clinical processes defining elements in the care of patients with COPD: smoking cessation counseling, influenza vaccination, motivation for physical activity, appropriate pharmacotherapy, patient education and collaborative care.

ELIGIBILITY:
Inclusion criteria:

* Males and females = 45yrs of age and
* Smoker or ex-smoker (with at least 10 PY) and
* Obstruction in spirometry FEV1/FVC< 0.7

Exclusion criteria:

* No obstruction in spirometry (FEV1/FVC > 0.7) or
* Patients with history of asthma or hay fever or
* Other concomitant pulmonary disease or
* Patients with malignancies of any other system and/or other severe disease with an estimated life expectancy of less than six months or
* Insufficient German language skills or
* Patients who contact the practice for emergencies only or as a substitute practice

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2013-09; Primary Completion 2017-01 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
"Quality of care process" | one year
  Difference in "quality of care process" (total increase in performed measures/fulfilled indicators) will be assessed after one year between COPD patients in the intervention and control group as reported by the patient

SECONDARY OUTCOMES:
Quality of life | one year
  We use the COPD Assessment Test (CAT). The CAT provides clinicians and patients with a reliable measure of overall COPD-related health status for the assessment and long-term follow-up of individual patients. The CAT is a validated short and simple patient-completed questionnaire that has been developed for use in routine clinical practice to measure the health status and grading the impact of COPD on patients' life. The CAT has very similar discriminative properties to the much more complex SGRQ (St. Georges Respiratory Questionnaire), and is available in different languages. It compromises 8 simple questions, 8 items on a scale 0-5 with a total scoring range of 0-40. CAT score <10 low impact, 10-20 medium impact >30 very high impact of COPD on patients life

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Rosemann, Prof MD, Principal Investigator — University Hospital Zurich, Institute of General Practice
Locations (1):
- Institute of General Practice, University of Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Steurer-Stey C, Markun S, Lana KD, Frei A, Held U, Wensing M, Rosemann T. The improving care in chronic obstructive lung disease study: CAROL improving processes of care and quality of life of COPD patients in primary care: study protocol for a randomized controlled trial. Trials. 2014 Mar 27;15:96. doi: 10.1186/1745-6215-15-96. PMID 24670200